CLINICAL TRIAL: NCT05160532
Title: Intraarticular Dextrose Prolotherapy for Symptomatic Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David C. Patchett, DO, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-008778
Record Dates: First submitted 2021-12-02; First posted 2021-12-16 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Four injections of placebo (Placebo Comparator): Subjects will receive four placebo intraarticular knee injections under ultrasound guidance. A placebo looks exactly like the study drug, but it contains no active ingredient.
  Interventions: Drug: Placebo
- One injection of DPT and three injections of placebo (Experimental): Subjects will receive one intraarticular knee injection under ultrasound guidance of dextrose prolotherapy (DPT), followed by three intraarticular knee injections of placebo under ultrasound guidance.
  Interventions: Drug: Placebo; Drug: Dextrose prolotherapy (DPT)
- Two injections of DPT and two injections of placebo (Experimental): Subjects will receive two intraarticular knee injection under ultrasound guidance of dextrose prolotherapy (DPT), followed by two intraarticular knee injections of placebo under ultrasound guidance.
  Interventions: Drug: Placebo; Drug: Dextrose prolotherapy (DPT)
- Four injections of DPT (Experimental): Subjects will receive four intraarticular knee injection under ultrasound guidance of dextrose prolotherapy (DPT).
  Interventions: Drug: Dextrose prolotherapy (DPT)

INTERVENTIONS:
Drug: Placebo — 5ml of normal saline (NS)
  Arms: Four injections of placebo; One injection of DPT and three injections of placebo; Two injections of DPT and two injections of placebo
Drug: Dextrose prolotherapy (DPT) — 25% dextrose, mixing 2.5ml of sterile water and 2.5ml of 50% dextrose.
  Arms: Four injections of DPT; One injection of DPT and three injections of placebo; Two injections of DPT and two injections of placebo

SUMMARY:
The purpose of this research is to learn more about treating Symptomatic Knee Osteoarthritis (OA) with an ultrasound-guided hypertonic dextrose injection. Researchers would like to determine best practice for injection frequency and effectiveness of the dextrose injection for symptomatic knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee OA by clinical criteria (American College of Rheumatology).
* Identification of knee osteoarthritis by a radiologist on an existing knee radiograph obtained within 3 years of enrollment.
* Moderate to severe knee pain for at least 3 months, defined as a score of ≥ 4 (on a 0-10 point numeric rating scale) in response to the question "What is the average level of your left/right knee pain in the past 3 months?".

Exclusion Criteria:

* Pregnancy.
* Diabetes.
* Anticoagulation therapy.
* History of total knee replacement.
* Prior knee prolotherapy or other regenerative product.
* Any knee injection within 3 months.
* Inflammatory (RA, gout, pseudogout etc.) or postinfectious knee arthritis.
* Daily use of opioid medication.
* Allergy or intolerance to study medication, corn allergy.
* Body mass index (BMI) greater than 40 kg/m^2.
* Comorbidity severe enough to prevent participation in the study protocol.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 4 weeks, 8 weeks, 16 weeks, 26 weeks, and 52 weeks
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) disease-specific tool used to measure physical function, pain, and stiffness in individuals with knee OA. Total scores range from 0-100, with higher scores indicating worse outcome.

SECONDARY OUTCOMES:
Change in pain | Baseline, 4 weeks, 8 weeks, 16 weeks, 26 weeks, and 52 weeks
  Measured using a visual analogue scale with 0 = no pain and 10=worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: David Patchett, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No